CLINICAL TRIAL: NCT05285722
Title: Adaptation and Testing of Cognitive Behavioral Therapy Resource of Turkish Version of ''Message to Dentist'' to Reduce Dental Anxiety in Children
Brief Title: Testing of Cognitive Behavioral Therapy Resource of Turkish Version
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altinbas University (Other)
Responsible Party: Principal Investigator, Aliye Tugce Gurcan, Assist.Prof., Altinbas University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AltinbasU
Record Dates: First submitted 2022-02-04; First posted 2022-03-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Dental Anxiety
Keywords: dental anxiety; cognitive behavioral therapy; pediatric dentistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dental anxiety group (Other): Children,
  * Aged 5-15 years
  * Having dental anxiety but not having negative experiences during dental treatment in childhood or adolescence
  * Without any systemical and mental diasabilities
  * Who volunteered to participate in the study and whose parental consent was obtained.
  Interventions: Behavioral: Cognitive Behavioral Therapy form for dental anxiety

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy form for dental anxiety — Message to Dentist form

SUMMARY:
This study aimed to evaluate the cognitive behavioral therapy source of Turkish version of the 'message to dentist' (MTD) with children attending two dental settings.

DETAILED DESCRIPTION:
Children aged 5-16 years attending a dental faculty clinic and a private dental office were invited to complete the MTD form. Children were asked to report how worried they felt, their level of pain they anticipated and the actual level of pain they experienced on a scale of 1-10 (with 1 being the best outcome).

ELIGIBILITY:
Inclusion Criteria:

Having dental anxiety but not having negative experiences during dental treatment in childhood or adolescence

* Without any systemical and mental diasabilities
* Who volunteered to participate in the study and whose parental consent was obtained.

Exclusion Criteria:

* not have dental anxiety
* having any systemical or mental disability
* having negative experiences during dental treatment in childhood or adolescence
* and who did not volunteer to participate in the study and did not have parental consent for the study were excluded.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 262 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
clinic differences and dental anxiety | 6 month
  according to CBT form, it will be evaluated
worry type of participants | 6 month
  according to Cognitive Behavioral Therapy form, it will be evaluated
Gender anxiety differences | 6 month
  according to Cognitive Behavioral Therapy form, it will be evaluated

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Altinbas University, Faculty of Dentistry, Istanbul, Bakirkoy
  - Altinba University Faculty of Dentistry, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Porritt J, Rodd H, Morgan A, Williams C, Gupta E, Kirby J, Creswell C, Newton T, Stevens K, Baker S, Prasad S, Marshman Z. Development and Testing of a Cognitive Behavioral Therapy Resource for Children's Dental Anxiety. JDR Clin Trans Res. 2017 Jan;2(1):23-37. doi: 10.1177/2380084416673798. Epub 2016 Nov 1. PMID 28879243